CLINICAL TRIAL: NCT02905253
Title: A Three-part Single-center, Phase 1 Study to Assess the Tolerability, Safety, Pharmacokinetics (Including Food Interaction), and Pharmacodynamics of Ascending Single and Multiple Doses of AC-084 in Healthy Subjects and to Investigate the Pharmacokinetics of a Single Dose of AC-084 in Healthy CYP2C9 Poor Metabolizers
Brief Title: A Study to Evaluate if AC-084 is Safe, Its Fate in the Body as Well as Its Potential Effects on the Body in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been terminated due to difficulties in recruiting subjects into Part C. No safety concerns contributed to the termination of the study
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AC-084-101
Record Dates: First submitted 2016-08-31; First posted 2016-09-19 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- AC-084, single ascending dose (Part A) (Experimental): AC-084 administered at different single dose levels in a sequential manner, and in a maximum of 7 dose levels starting from 1 mg (number of cohorts and dose levels will depend on the safety and pharmacokinetic results of the previous cohort). Each dose level will be investigated in a new group of at least 8 healthy male subjects (6 on active drug and 2 on placebo)
  Interventions: Drug: AC-084
- Placebo,single ascending dose (Part A) (Placebo Comparator): Matched placebo administered as single ascending doses in parallel to AC-084
  Interventions: Drug: Placebo
- AC-084, multiple ascending dose (Part B) (Experimental): AC-084 administered in a twice daily (b.i.d.) dosing regimen at multiple dose levels. The starting dose will be between 1 and 30 mg and will be selected on the basis of the safety and pharmacokinetic results of the part A. Each dose level will be investigated in a new group of at least 8 healthy male subjects (6 on active drug and 2 on placebo)
  Interventions: Drug: AC-084
- Placebo,multiple ascending dose (Part B) (Placebo Comparator): Matched placebo administered as multiple ascending doses in parallel to AC-084
  Interventions: Drug: Placebo
- AC-084, single dose (Part C) (Experimental): Up to 6 subjects in part C will receive AC-084 administered at a single dose (foreseen to be 100 mg)
  Interventions: Drug: AC-084

INTERVENTIONS:
Drug: AC-084 — Hard gelatin capsules for oral administration formulated in strengths of 1 mg, 10 mg, and 100 mg
  Arms: AC-084, multiple ascending dose (Part B); AC-084, single ascending dose (Part A); AC-084, single dose (Part C)
Drug: Placebo — Placebo capsules matching AC-084 capsules
  Arms: Placebo,multiple ascending dose (Part B); Placebo,single ascending dose (Part A)

SUMMARY:
The primary purpose of this first-in-man study is to investigate whether AC-084 is safe and well-tolerated when orally administered at single- and multiple-ascending dose to healthy adults

DETAILED DESCRIPTION:
The study is designed in three parts, A, B and C

Part A: single-center, double-blind, randomized, placebo-controlled, single ascending dose

Part B: single-center, double-blind, randomized, placebo-controlled, multiple ascending dose

Part C: single-center, open-label, single dose in CYP2C9 poor metabolizers

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure
* Healthy male subjects for Part A, healthy male and female subjects for Part B and Part C aged between 18 and 55 years (inclusive) at screening
* No clinically significant findings on physical examination at screening
* Body mass index (BMI) of 18.0 to 28.0 kg/m2 (inclusive) at screening
* CYP2C9 poor metabolizers (Part C)

Exclusion Criteria:

* History or clinical evidence of any disease and/or existence of any surgical or medical condition that might interfere with the absorption, distribution, metabolism or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions
* Treatment or substances known to induce CYP enzyme drug metabolism within 30 days prior to first study treatment administration
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol
* Known allergic reactions or hypersensitivity to the study treatment or drugs of the same class, or any of their excipients
* For Part A and Part B, CYP2C9 poor metabolizers enrolled in a cohort to be dosed with single or multiple dose of 500 mg or higher of ACT-774312 (confirmed by genotyping before enrollment)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) (Part A) | From dosing until day 4
  Treatment-emergent AEs and treatment-emergent serious AEs
Number of participants with adverse events (AEs) (Part B) | From dosing until day 8
  Treatment-emergent AEs and treatment-emergent serious AEs
Number of participants with adverse events (AEs) (Part C) | From dosing until day 6
  Treatment-emergent AEs and treatment-emergent serious AEs
Incidence of safety events of interest (Part A) | From dosing until day 4
  Events of interest are any abnormalities in ECG, vital signs or laboratory test results
Incidence of safety events of interest (Part B) | From dosing until day 8
  Events of interest are any abnormalities in ECG, vital signs or laboratory test results
Incidence of safety events of interest (Part C) | From dosing until day 6
  Events of interest are any abnormalities in ECG, vital signs or laboratory test results

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) following single oral ascending doses (Part A) | From dosing until day 4
  Cmax is derived from the observed plasma concentration-time curves
Maximum plasma concentration (Cmax) following single oral ascending doses (Part B) | From dosing until day 8
  Cmax is derived from the observed plasma concentration-time curves
Maximum plasma concentration (Cmax) following single oral ascending doses (Part C) | From dosing until day 6
  Cmax is derived from the observed plasma concentration-time curves
Time to reach Cmax (tmax) following single oral ascending doses (Part A) | From dosing until day 4
  Tmax is derived from the observed plasma concentration-time curves
Time to reach Cmax (tmax) following single oral ascending doses (Part B) | From dosing until day 8
  Tmax is derived from the observed plasma concentration-time curves
Time to reach Cmax (tmax) following single oral ascending doses (Part C) | From dosing until day 6
  Tmax is derived from the observed plasma concentration-time curves
Terminal half-life [t(1/2)] following single oral ascending doses (Part A) | From dosing until day 4
Terminal half-life [t(1/2)] following single oral ascending doses (Part B) | From dosing until day 8
Terminal half-life [t(1/2)] following single oral ascending doses (Part C) | From dosing until day 6
Area under the plasma concentration-time curve (AUC) following single oral ascending doses (Part A) | From dosing until day 4
  AUC is defined for the time intervals from zero to time t of the last measured concentration above the limit of quantification and from zero to infinity
Area under the plasma concentration-time curve (AUC) following single oral ascending doses (Part B) | From dosing until day 8
  AUC is defined for the time intervals from zero to time t of the last measured concentration above the limit of quantification and from zero to infinity
Area under the plasma concentration-time curve (AUC) following single oral ascending doses (Part C) | From dosing until day 6
  AUC is defined for the time intervals from zero to time t of the last measured concentration above the limit of quantification and from zero to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Martine Géhin, PhD, Study Director — Actelion
Locations (1):
- Covance Clinical Research Unit, Leeds, United Kingdom